CLINICAL TRIAL: NCT05006391
Title: Tele-Coaching CBE Study: Evaluating the Implementation of an Online Community-Based Exercise (CBE) Intervention Using Tele-Coaching to Enhance Physical Activity Among Adults Living With HIV
Brief Title: Tele-Coaching Community-Based Exercise (CBE) Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: YMCA (Other); Ontario HIV Treatment Network (Network)
Responsible Party: Principal Investigator, Kelly O'Brien, Associate Professor, University of Toronto
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: REB Protocol #40410
Record Dates: First submitted 2021-07-21; First posted 2021-08-16 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2023-05

CONDITIONS: Hiv
Keywords: HIV; exercise; community-based exercise; tele-rehabilitation; tele-health; rehabilitation; disability; tele-coaching
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tele-Coaching (Online) Community-Based Exercise (Experimental): This study involves two phases: a six month online Community-Based Exercise Intervention (Phase 1), followed by a six month Follow-Up Monitoring Phase (Phase 2).
  Interventions: Other: Tele-Coaching (Online) Community-Based Exercise

INTERVENTIONS:
Other: Tele-Coaching (Online) Community-Based Exercise — PHASE 1-Intervention Phase (6 months): Participants will engage in an individual tailored home-based exercise program involving aerobic, resistance, balance and flexibility training ~60min, 3 times per week for 24 weeks. Intervention will include: Component 1) biweekly 60 min personal online coaching with a certified trainer from the YMCA (13 sessions) who will monitor and progress exercise intensity; Component 2) weekly online group-based exercise classes ~60 min each led by a trainer at YMCA; Component 3) monthly online evidence-based self-management education sessions focused on topics related to self-management and health, and physical activity living with HIV; and Component 4) a wireless physical activity monitor (WPAM) to self-monitor steps, distance, calories burned, and active minutes.
  PHASE 2: Post-Intervention (6 months): Participants will be encouraged to continue with unsupervised home / outdoor-based exercise 3 times per week and to continue using their WPAM throughout.

SUMMARY:
The primary aim of this research is to evaluate the implementation of an online tele-coaching community-based exercise (CBE) intervention with adults living with HIV.

DETAILED DESCRIPTION:
Investigators will use the RE-AIM (Reach-Effectiveness-Adoption-Implementation-Maintenance) Framework to evaluate the tele-coaching CBE intervention. The RE-AIM Framework includes criteria to evaluate the impact and translation of an intervention at both individual and organizational levels in order to promote uptake, transferability and ultimate enhance the impact of health promotion interventions.

Specific study objectives are: 1) To determine the extent (proportion of sessions attended, frequency, intensity, time, type) to which adults living with HIV participate in the intervention (Reach); 2) To assess the impact of the intervention on physical activity, health, and engagement in the care cascade (Effectiveness); 3) To assess engagement in exercise for adults living with HIV over time (physical activity, adherence) (Maintenance); and 4) To evaluate the a) process (strengths, challenges, accessibility, cost, fidelity) and b) feasibility of sustainability of the implementation, from the perspective of adults living with HIV, representatives of community-based organizations (CBOs), health and fitness centres, health providers, and policy stakeholders to build capacity, products, and considerations for broader implementation (Implementation and Adoption).

Investigators will conduct a prospective longitudinal mixed methods intervention study to evaluate the implementation of an innovative online tele-coaching CBE intervention with adults living with HIV. They will use a combination of quantitative (self-reported questionnaires, fitness assessments) to assess outcomes bimonthly during the tele-coaching CBE intervention (6 months) and during a follow-up monitoring phase (6 months) to evaluate the short and long term impact of online CBE. Investigators will use a qualitative longitudinal design using interviews to assess processes and outcomes at baseline (0 months), post-intervention (6 months) and post-follow-up (12 months).

ELIGIBILITY:
Inclusion Criteria:

* Adults (18 years and older) living with HIV who consider themselves medically stable and safe to engage in exercise.
* Access to technology (computer/tablet, Wi-Fi, web-cam).
* Willing to take part in a 12 month study involving thrice weekly exercise.

Exclusion Criteria:

• Not applicable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2021-05-17 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Physical Activity | Weekly outcome assessment throughout the intervention phase (6 months) and follow-up monitoring phase (6 months) for a total of 12 months (48 weeks).
  Change in trend (slope) in self-reported physical activity during the intervention phase (6 months) and the follow-up phase (6 months) as measured by i) whether they achieved the weekly recommended Canadian Physical Activity Guidelines, and ii) the number of days in the past week engaged in ≥30 min of moderate to vigorous physical activity (single item physical activity questionnaire).

SECONDARY OUTCOMES:
Disability | Bimonthly outcome assessment throughout the intervention phase (6 months) and follow-up monitoring phase (6 months) for a total of 13 time points.
  Change in trend (slope) in disability as during the intervention phase (6 months) and the follow-up phase (6 months) as measured by the Short Form HIV Disability Questionnaire (SF-HDQ).
Health | Bimonthly outcome assessment throughout the intervention phase (6 months) and follow-up monitoring phase (6 months) for a total of 13 time points.
  Change in trend (slope) in disability as during the intervention phase (6 months) and the follow-up phase (6 months) as measured by the EQ-5D-5L.
Mental Health | Bimonthly outcome assessment throughout the intervention phase (6 months) and follow-up monitoring phase (6 months) for a total of 13 time points.
  Change in trend (slope) in disability as during the intervention phase (6 months) and the follow-up phase (6 months) as measured by the Patient Health Questionnaire (PHQ-8).
Engagement in Care | Bimonthly outcome assessment throughout the intervention phase (6 months) and follow-up monitoring phase (6 months) for a total of 13 time points.
  Change in trend (slope) in disability as during the intervention phase (6 months) and the follow-up phase (6 months) as measured by the HIV Index of Engagement questionnaire.

OTHER OUTCOMES:
Extrinsic Contextual Factor - HIV Stigma | Bimonthly outcome assessment throughout the intervention phase (6 months) and follow-up monitoring phase (6 months) for a total of 13 time points.
  Change in trend (slope) in disability as during the intervention phase (6 months) and the follow-up phase (6 months) as measured by the Short Form HIV Stigma Scale.
Intrinsic Contextual Factor - Mastery | Bimonthly outcome assessment throughout the intervention phase (6 months) and follow-up monitoring phase (6 months) for a total of 13 time points.
  Change in trend (slope) in disability as during the intervention phase (6 months) and the follow-up phase (6 months) as measured by the Pearlin Mastery Scale.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Toronto, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Data Availability Statement: Data are available upon reasonable request. Members of the research team will have access to an anonymized aggregated dataset for this study. An aggregated dataset for the study will be made available upon reasonable request to the corresponding author in accordance with the Research Ethics Board requirements of the University of Toronto.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data sharing may occur within 5 years from study completion as this is the timeframe outlined in the Research Ethics Board (REB) approval, after which the data will be destroyed.
Access Criteria: Data are available upon reasonable request. An aggregated dataset for the study will be made available upon reasonable request to the corresponding author in accordance with the Research Ethics Board requirements of the University of Toronto. The request should include the research objectives in which the team is requesting use of the data, details of the team / individuals requesting the data, the variables requested, and any funding to support.

REFERENCES:
- [Derived] Ibanez-Carrasco F, McDuff K, Da Silva G, Bayoumi AM, Chan Carusone S, Loutfy M, Tang A, Ahluwalia P, Avery L, O'Brien KK. Qualitative insights from an online community-based exercise intervention for persons living with HIV. Front Rehabil Sci. 2025 Aug 25;6:1602007. doi: 10.3389/fresc.2025.1602007. eCollection 2025. PMID 40927745
- [Derived] Su TT, Chan Carusone S, McDuff K, Ibanez-Carrasco F, Tang A, Bayoumi AM, Loutfy M, Avery L, Da Silva G, Furlan A, Trent H, Ilic I, Pandovski Z, Zobeiry M, Ahluwalia P, Krizmancic K, Jiancaro T, Torres B, Solomon P, O'Brien KK. Goals in motion: exploring goal setting among adults living with HIV who participated in an online community-based exercise intervention. Front Rehabil Sci. 2025 Jul 31;6:1644139. doi: 10.3389/fresc.2025.1644139. eCollection 2025. PMID 40820990
- [Derived] O'Brien KK, Ibanez-Carrasco F, Carusone SC, Bayoumi AM, Tang A, McDuff K, Jiancaro T, Da Silva G, Torres B, Loutfy MR, Islam S, Lindsay J, Price C, Zobeiry M, Pandovski Z, Illic I, Ahluwalia P, Brown DA, Avery L, Solomon P. Piloting an online telecoaching community-based exercise intervention with adults living with HIV: protocol for a mixed-methods implementation science study. BMJ Open. 2023 Mar 30;13(3):e067703. doi: 10.1136/bmjopen-2022-067703. PMID 36997255